CLINICAL TRIAL: NCT01505504
Title: Mirtazapine in Alzheimer-associated Weight Loss: a Retrospective Phase IV Study
Brief Title: Mirtazapine in Alzheimer-associated Weight Loss
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Kurt Segers, Principal Investigator, Brugmann University Hospital
Other Study IDs: MIRTA-2012
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Alzheimer's Disease; Weight Loss; Mixed Dementia; Dementia
MeSH Terms: conditions — Alzheimer Disease; Weight Loss; Mixed Dementias; Dementia | interventions — Mirtazapine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: mirtazapine — 30 mg at bedtime
  Other Names: Remergon

SUMMARY:
Weight loss is a frequent problem associated with Alzheimers disease (AD). Mirtazapine has weight loss as a frequent side effect.

The aim of this retrospective study is to check whether mirtazapine 30 mg (once daily) can counteract weight loss in patients with AD or mixed dementia (AD + vascular).

ELIGIBILITY:
Inclusion Criteria:

* AD or mixed dementia
* documented weight loss
* mirtazapine 30 mg explicitly prescribed against weight loss

Exclusion Criteria:

* no treatment compliance
* other causes of weight loss
* other interventions against weight loss

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with established diagnosis of AD or mixed dementia with reported weight loss
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2004-01; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
body weight | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brugmann, Brussels, Belgium